CLINICAL TRIAL: NCT06011486
Title: Expansion of Virus-Specific Lymphocytes for Cell Therapy in Immunosuppressed Patients Who Underwent Bone Marrow Transplantation.
Brief Title: Expansion of Virus-Specific Lymphocytes for Cell Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1226-7367
Record Dates: First submitted 2023-06-16; First posted 2023-08-25 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: CMV Viremia; CMV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphocyte infusion (Experimental): Patients with CMV disease or reactivation will be included for receiving donor-CMV-specific cells
  Interventions: Combination Product: Lymphocyte infusion (ImmuneCellVir-I)

INTERVENTIONS:
Combination Product: Lymphocyte infusion (ImmuneCellVir-I) — Infusion of donor CMV specific cells into patients eligible to the trial
  Other Names: CMV-specific cells infusion

SUMMARY:
Infections and reactivation of human cytomegalovirus (CMV), adenovirus, Epstein-barr and polyoma virus infections are frequent causes of morbidity and mortality and are a source of serious complications in patients undergoing allogeneic bone marrow transplantation.

In this project we will prepare specific T lymphocytes from blood donor, select cells CMV-specific by interferon gamma capture and treat patients with CMV viral infections. These cells will be used as antiviral therapy in transplanted patients whom do not respond to conventional therapies or in patients whose conventional therapy may be toxic in the context of transplantation. In this context, CMV reactivation can lead to serious complications in patients, such as irreversible neurological changes, pulmonary, gastrointestinal and ophthalmologic complications, among others, in addition to prolonged hospitalizations, leading to significant morbidity and mortality , both in the health sector public as private.

This project may represent an important therapeutic modality using cell of the shelf as a source of therapy for different patients and contributing to reduced morbidity / mortality after transplantation, as well as a reduction in the hospitalization period.

DETAILED DESCRIPTION:
The proposed clinical trial is a phase I single-arm infusion study of cytomegalovirus (CMV)-specific lymphocytes derived from buffy-coat derivatives of platelet donors (ImmuneCellVir-I). T lymphocytes are expanded, stimulated with peptide (pp65) from the viral capsid and selected according to interferon-γ (INF-γ) production in response to the stimulus. After selection, the lymphocytes will be frozen and released for infusion into recipients according to HLA compatibility, result of aerobic/anaerobic cultures and special microorganisms/fungi, endotoxin, donor serological assays, PCR for CMV, EBV and B19 of the product, NAT HCV, HIV, HBS and HTLV-1/2 of the product, and results of impurity and potency tests of the product.

The main objective of the study is to evaluate the safety and tolerability of Cytomegalovirus (CMV)-specific Lymphocyte infusion in patients with CMV infection who do not respond to conventional therapies or whose pharmacological therapy may be toxic in the post-transplant context. As secondary outcome to determine the effectiveness of the infusion of CMV-specific lymphocytes The main benefit to potential participants is the treatment of cytomegalovirus infection for patients who are refractory or intolerant to the established drug treatment. Furthermore, the infusion of CMV-specific lymphocytes could potentially help in the immune reconstitution of patients. The expectation is that, with this therapeutic modality, it will be possible to treat patients who have no other treatment alternative. While, the known possible risks are related to cryopreserved allogeneic product infusion reactions and potential risk of graft versus host disease.

The possible mechanism of action of this therapy would be through the infused CMV-specific donor cells that would recognize the CMV-infected cells in the patient. CD4 T lymphocytes amplify the immune response by secreting cytokines, CD8 T lymphocytes attack CMV-infected cells, releasing perforins and granzymes.

Cytomegalovirus (CMV)-specific lymphocytes will be administered intravenously. Patients will receive therapy containing a total amount of 1x106 CMV-specific T lymphocytes, equivalent to a 1-2x104 dose/kg of recipient weight, which can be repeated on up to 2 occasions with a minimum interval of 2 weeks between infusions, if the patient persists with the presence of inclusion criteria in the study. The trial will be performed in accordance with protocol, good clinical practice and regulatory requirements.

At this time, it is not possible to state that all research participants will benefit directly from this study. However, its development will allow a better knowledge of this cellular therapy, allowing an improvement of the protocol and greater efficiency in future protocols to be carried out. It is expected that the proposed treatment generates at least a better quality of life for research participants, with a decrease in complications resulting from the disease.

Infusion reactions, development of graft versus host disease (GvHD) and Immunogenicity The primary outcomes of safety of ImmuneCellvir -I will be verified in the patients that will be followed during infusion and 7 consecutive weeks after infusion, and also 100, 180 and 365 days. After cell infusion, patients will be monitored for vital signs (mmHg), pulse rate and blood oxygen level every 15 minutes and must be instructed to contact the study team for any unusual symptoms. After infusion, will be 6 visits (1/week) and 100 days, 6 months and 1 year, after infusion. Patients will be followed for clinical signs and symptoms of acute and chronic GvHD , as gastrointestinal tract alterations, skin, eye, liver, musculoskeletal and lung changes. Patient will be tested for 7 weeks for Bilirubin (μmol/L), Alkaline phosphatase (U/L), Gamma-glutamyl Transferase (U/L) , glutamic-oxaloacetic transaminase/ glutamic pyruvic transaminase (U/L), blood cells count (cells/mm3), creatinine (mg/dL), urea(mg/dL), Serum level of tacrolimus/cyclosporine (mg/dL). For Immunogenicity will be measured the development of anti Human Leukocyte Antigen antibodies in the patient.

The secondary outcome will be measured by the evaluation of clinical symptoms score, level of CMV copies and anti-CMV response. The secondary or exploratory outcome will be performed for as indicative of efficacy. This outcome will be reported as a score of clinical symptoms, comparing the symptoms before and after the infusion. Laboratorial tests will be performed for 7 consecutive weeks after the infusion to demonstrated the patient clinical improvement as the rate of CMV viral load (copies/mL), rate of anti-CMV response in the peripheral blood of patients by ELISpot (IFN-y spots/10x6cells). The patients can be also evaluated for specific exams (if required) depend on the site of infection as computed tomography, colonoscopy, eye fundus examination and biopsy. In addition, assays to determine cell biodistribution as chimerism (%) after infusion will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide signed informed consent.
* Must be between 18 and 75 years old at the time of signing the consent form
* Having undergone allogeneic hematopoietic stem cell transplantation (related, unrelated, haploidentical or cord blood transplant)
* Negative pregnancy test for women of childbearing age (non-fertile age defined as post-menopausal over one year, or surgically sterilized); Acceptance of the use of contraceptive methods by sexually active men and women of childbearing age;
* Present with clinically significant CMV infection and one of the following conditions:
* Refractory CMV infection, defined as over a 1log increase in blood or plasma CMV copies number after 2 weeks of treatment with appropriate anti-CMV medication (treatment with ganciclovir, valganciclovir, or foscarnet)
* Probable refractory CMV infection, defined as persistence of CMV DNA in blood or plasma at the same level or under 1 log increase after 2 weeks of treatment with appropriate anti-CMV medication (treatment with ganciclovir, valganciclovir, or foscarnet)
* Presence of resistant CMV, defined by the presence of a known genetic mutation that reduces susceptibility to one or more antiviral medications
* Refractory CMV disease, defined as worsening of signs and symptoms and/or progression to CMV disease after 2 weeks of appropriate antiviral therapy
* Restrictions or complications related to conventional therapy, which make it impossible to carry out conventional drug treatment defined as cytopenias with neutrophils under 1000 per microliter, platelets under 100,000 per microliter related to the use of ganciclovir or valganciclovir and nephrotoxicity with an increase of 1.5 times in the baseline creatinine with the use of foscavir.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients who do not agree to participate in the study or sign the consent form
* Patients reporting allergy to murine antibodies or iron-dextran
* Patients with grade 3 or 4 graft versus host disease/graft versus host disease in activity/treatment
* Pregnant or lactating patients
* Patients with uncontrolled bacterial and/or fungal infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with immediate infusion reactions | 3 hours
  Safety of cytotoxic T cell (CTL) based on patients with grade 3 immediate adverse events that are at least possibly related to the CTL infusion within 3 hours of the CTL infusion, using the grade as follows: Grade 1 Mild; asymptomatic or mild symptoms. Grade 2 Moderate symptoms. Grade 3 Severe with Life-threatening consequences.
Development of Acute graft versus host disease (GvHD) | 6 weeks
  Number of Patients that present Acute GvHD Grades III-IV [ Time Frame: 6 weeks] Safety of cytotoxic T Cell (CTL) will be based on patients with acute GvHD grades III-IV within 6 weeks after the last dose of CTL. Acute GVHD grading will be performed according to NIH criteria (1). Grade 0 represents no acute GvHD. Grade 4 represents the most severe acute GvHD.
  1-Harris AC, Young R, Devine S, Hogan WJ, Ayuk F, et al. International, Multicenter Standardization of Acute Graft-versus-Host Disease Clinical Data Collection: A Report from the Mount Sinai Acute GVHD International Consortium. Biol Blood Marrow Transplant. 2016;22(1):4-10.
Development of Non-Hematological Adverse events | 6 weeks
  Number of Patients With Grades 3 Non-hematologic Adverse Events Related to the T Cell Product [ Time Frame: 6 weeks ] Safety of VSTs based on patients with grade 3 non-hematologic adverse events that are at least possibly related to the CTL infusion within 6 weeks of the last CTL dose, using the grade as follows: Grade 1 Mild; asymptomatic or mild symptoms. Grade 2 Moderate symptoms. Grade 3 Severe with Life-threatening consequences.
Risk for chronic GVHD [ Time Frame: At 6 and12 months post CTL infusion ] | 6 to 12 montas
  Survival analysis method will be applied. Time to chronic GVHD will be defined from time of the last CTL infusion to the onset of chronic GVHD, or the last clinical assessment date if no chronic GVHD. Cumulative incidence of chronic GVHD at 6 and 12 months will be estimated.

SECONDARY OUTCOMES:
Antiviral activity defined as response to viral load [ Time Frame: 6 weeks ] | 6 weeks
  Complete response, partial , or no response will be defined and proportion of each outcome will be calculated.
Rate of anti-CMV response improvement in the peripheral blood of participants [ Time Frame: 6 weeks ] | 6 weeks
  Anti-CMV response will be measured by ELISpot (IFN-y spots/10e6 cells)
Clinical response to CTL infusions [ Time Frame: At 6 weeks and 3 months ] | 6 weeks and 3 month
  In cases with CMV disease, clinical response can be evaluated with evaluation of the involved organ with specific exams (if required) as computed tomography, colonoscopy, eye fundus examination and biopsy .

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Hamerschlak, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil